CLINICAL TRIAL: NCT01245647
Title: Pharmacotherapy for Hazardous Drinking in HIV Infected Women: Randomized Trial
Brief Title: Will Having Alcohol Treatment Improve Functioning?
Acronym: WHAT-IF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AA018934-01-N; R01AA018934-01 (NIH)
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Results first posted 2014-02-27 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-04

CONDITIONS: HIV; Alcoholism
Keywords: women; HIV; alcohol; medication; adherence; acceptability
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar Pill, 50mg, once per day for 4 months (Placebo Comparator): Placebo: One third of the participants will receive placebo pills that look the same as the active comparator but are really just inert pills. Each study participant will take a single pill once a day for 4 months.
  Interventions: Other: Sugar pill, 50mg, once per day for 4 months
- Naltrexone, 50mg, once per day for 4 months (Active Comparator): Naltrexone: Two thirds of the total study participants will receive the medication naltrexone. Each study participant will take a single pill once a day for 4 months.
  Interventions: Drug: Naltrexone, 50mg, once per day for 4 months

INTERVENTIONS:
Drug: Naltrexone, 50mg, once per day for 4 months — Naltrexone: Two thirds of the total study participants will receive the medication naltrexone. Each study participant will take a single pill once a day for 4 months.
  Other Names: Naltrexone
  Arms: Naltrexone, 50mg, once per day for 4 months
Other: Sugar pill, 50mg, once per day for 4 months — Placebo: One third of the participants will receive placebo pills that look the same as the active comparator but are really just inert pills. Each study participant will take a single pill once a day for 4 months.
  Other Names: Inert sugar pill
  Arms: Sugar Pill, 50mg, once per day for 4 months

SUMMARY:
The purpose of the study is to find out if a medication,naltrexone is helpful for HIV-infected women who sometimes drink too much. The study will try to find out whether women like the medication, whether the medication helps them cut back on their drinking, and whether it helps improve their overall health. Naltrexone has not been used widely among people who are engaged in less severe drinking and in primary health care settings. Therefore, the investigators would like to determine whether it is helpful among women who sometimes drink 4 or more drinks per occasion or 7 or more drinks per week. The investigators hypothesize that by taking naltrexone, women with hazardous drinking pattern will reduce their drinking which in turn will improve their medication adherence, improve their health and quality of life.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the acceptability and effectiveness of a treatment program for hazardous drinking, delivered within HIV-clinic outpatient settings, that involves oral naltrexone. The central hypothesis is that women randomized to the treatment program will have decreased rates of hazardous drinking and improved clinical and behavioral health outcomes that are associated with hazardous drinking. The investigators have formulated this hypotheses based on the existing literature, the preliminary data and the clinical experience. The investigators hypothesize that women randomized to receive an alcohol treatment intervention will be less likely to have hazardous drinking behavior 6-months after enrollment, compared to women who received similar assessments but no formal treatment intervention. The investigators hypothesize that 4-months after enrollment, women randomized to receive an alcohol treatment intervention will have improved adherence to HIV antiretroviral therapy, improved CD4 cell counts, reduced HIV viral load, and reduced risky sexual behavior, compared to women who receive similar assessments but no formal intervention.

The investigators will recruit 90 women from 3 different sites in Florida, Washington DC and Chicago. Of those 90 women 60 will receive naltrexone and 30 will receive placebo. Study participants will take the medication for 4 months but the investigators will follow them for 7 months. At baseline, 2 months, 4 months and 7 months, the investigators will administer study questionnaires and assess their liver enzymes, CD4 count and viral load. The investigators will also follow them up at month 1 and 3 to reinforce the medication intake and to assess for any possible side effects.

New treatment options are available, but their impact on hazardous drinking has not yet been evaluated among HIV-infected women, many of whom are poor, minorities, or who have associated mental health or substance abuse problems. Delivery of therapeutic interventions must be improved in order to reduce hazardous drinking in women with HIV/AIDS. The proposed research is significant because the therapy will be offered within HIV clinic settings and will potentially improve the health of a population that is significantly undertreated. In addition to determining the effectiveness of an alcohol treatment intervention, the investigators will also identify key barriers and facilitators associated with adherence to pharmacologic treatment for alcohol in women with hazardous drinking. The findings will directly impact the type and quality of care for hazardous drinking in this subset of HIV-infected individuals and will inform both primary and secondary prevention efforts

ELIGIBILITY:
Inclusion Criteria:

* Hazardous drinking: defined by the NIAAA as either of the following:

  1. binge drinking (4 or more drinks per occasion at least twice monthly), (NIAAA 2005) - OR
  2. high quantity-frequency (>7 or drinks per week)
* Age 18 or over
* Female
* HIV-infected documented by a rapid HIV test or any licensed ELISA test kit and confirmed by a repeat ELISA, Western Blot, HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA viral load or a second antibody test by a method other than ELISA at any time prior to study entry.
* Able to understand and comply with planned study procedures.
* Willing and able to provide informed consent.

Exclusion Criteria:

* Contraindications to treatment with naltrexone: current physiologic opiate dependence; current daily prescription opioid medications; positive urine drug test for opioids; allergic to naltrexone; significantly abnormal baseline liver enzymes (AST or ALT ≥ 5 times normal); on dialysis for renal failure
* currently taking oral medications for tuberculosis.
* Currently pregnant or positive pregnancy test.
* currently breastfeeding.
* Currently taking an alcohol treatment medication (disulfiram, topiramate, naltrexone, acamprosate).
* currently homeless, unable to provide mailing address, or has plans to move from area within next 7 months.
* Unable to communicate in English.
* Research coordinator assessment that participant cannot comprehend the study or consent procedures
* Has current prognosis of less than 1 year to live
* Abnormal vital signs at enrollment visit
* Currently on treatment for Hepatitis C (HCV) infection
* Prisoner status

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Cook, MD, MPH, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - Women's Interagency HIV Study, Washington D.C., District of Columbia
  - University of Florida Health Science Center, Jacksonville, Florida
  - Women's Interagency HIV Study, Chicago, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited participants from 3 sites in 3 cities: Washington, D.C., Chicago, and Jacksonville from December 2010 to February 2012. The last participant completed her 7-Month follow-up at October 2012.
Groups:
- Sugar Pill, 50mg, Once a Day for 4 Months.: Placebo: placebo pills looked the same as the active comparator but were really sugar pills. Each study participant in this arm took a single pill once a day for 4 months.
- Naltrexone, 50mg, Once a Day for 4 Months: Naltrexone 50mg pills (single oral capsule): Each study participant in this arm took a single pill once a day for 4 months.
Period: Overall Study
Arm/Group | Sugar Pill, 50mg, Once a Day for 4 Months. | Naltrexone, 50mg, Once a Day for 4 Months
Started | 7 | 12
Completed | 7 | 8
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill, 50mg, Once a Day for 4 Months | Naltrexone, 50mg, Once a Day for 4 Months | Total
Number analyzed (Participants) | 7 | 12 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 12 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (9.3) | 48.7 (6.6) | 49.3 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 19
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 12 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Drinks Per Week
Description: Average number of standard alcohol drinks per week, as measured by timeline follow-back. A drink typically contains about 0.6 grams of alcohol, and generally represents 1 12-oz beer, 1 5-oz glass of wine, or one shot of liquor.
Time Frame: Month 4
Population: All participants who provided data at the 4-month follow-up were included (n=15), which is 79% of persons who were randomized.
Measure: Mean (Standard Deviation); unit: standard alcohol drinks per week
Arm/Group | Sugar Pill, 50mg, Once a Day for 4 Months. | Naltrexone, 50mg, Once a Day for 4 Months
Number analyzed (Participants) | 7 | 8
standard alcohol drinks per week | 13.8 (12.4) [0.7 to 14.1] | 12.0 (16.5) [-2.6 to 5.3]
Statistical Analysis 1: Comparison: Sugar Pill, 50mg, Once a Day for 4 Months. vs Naltrexone, 50mg, Once a Day for 4 Months; Test type: Superiority or Other; p = 0.82, t-test, 2 sided

2. Secondary Outcome: HIV Medication Adherence (95% or Better)
Description: Medication adherence was measured on a visual analogue scale ranging from 0 - 100, and indicating what percentage of the persons' HIV medication was taken on schedule over the past week (self-report). A score of 95% or better was considered adherent, and we report the proportion of persons who were adherent in each group.
Time Frame: Month 4
Population: Only persons who reported current HIV medication use (n=13) were considered for this outcome, and we included data from the 12 persons who completed the 4-month assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Sugar Pill, 50mg, Once a Day for 4 Months. | Naltrexone, 50mg, Once a Day for 4 Months
Number analyzed (Participants) | 6 | 6
percentage of participants | 50 | 50
Statistical Analysis 1: Comparison: Sugar Pill, 50mg, Once a Day for 4 Months. vs Naltrexone, 50mg, Once a Day for 4 Months; Test type: Superiority or Other; p = 1.0, Fisher Exact

3. Secondary Outcome: Risky Sexual Behaviors
Description: Risky sexual behavior was a dichotomous outcome for each participant at each time point, defined as having any non-condom-protected sex with a males who have an unknown/negative HIV status in the previous 30 days.
Time Frame: 4 months
Measure: Number; unit: percentage of persons with risky sex
Arm/Group | Sugar Pill, 50mg, Once a Day for 4 Months. | Naltrexone, 50mg, Once a Day for 4 Months
Number analyzed (Participants) | 7 | 7
percentage of persons with risky sex | 0 | 29
Statistical Analysis 1: Comparison: Sugar Pill, 50mg, Once a Day for 4 Months. vs Naltrexone, 50mg, Once a Day for 4 Months; Test type: Superiority or Other; p = 0.46, Fisher Exact

4. Secondary Outcome: HIV Viral Load Suppressed
Description: Viral load was classified as either suppressed (HIV viral load <50 copies/ml) or not suppressed (HIV viral load >50 copies/ml). We report the proportion of participants who had a suppressed viral load (higher number is better)
Time Frame: 4 months
Measure: Number; unit: percentage of persons with suppressed VL
Arm/Group | Sugar Pill, 50mg, Once a Day for 4 Months. | Naltrexone, 50mg, Once a Day for 4 Months
Number analyzed (Participants) | 7 | 8
percentage of persons with suppressed VL | 43 | 88
Statistical Analysis 1: Comparison: Sugar Pill, 50mg, Once a Day for 4 Months. vs Naltrexone, 50mg, Once a Day for 4 Months; Test type: Superiority or Other; p = 0.12, Fisher Exact — no significant difference by Fisher exact test

5. Secondary Outcome: CD4 Count (Mean)
Description: Results from CD4 cell count result obtained either as lab specifically for this study, or from lab results that were collected at the same time point for a different study or clinical indication.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: CD4 count (cells/ml)
Arm/Group | Sugar Pill, 50mg, Once a Day for 4 Months. | Naltrexone, 50mg, Once a Day for 4 Months
Number analyzed (Participants) | 6 | 7
CD4 count (cells/ml) | 669 (478) | 761 (207)
Statistical Analysis 1: Comparison: Sugar Pill, 50mg, Once a Day for 4 Months. vs Naltrexone, 50mg, Once a Day for 4 Months; Test type: Superiority or Other; p = 0.67, t-test, 2 sided

ADVERSE EVENTS:
Groups:
- Sugar Pill, 50 mg Once a Day for 4 Months: Placebo: placebo pills looked the same as the active comparator but were really sugar pills. Each study participant in this arm took a single pill once a day for 4 months.
- Naltrexone, 50mg Pill Once a Day for 4 Months: Naltrexone 50mg pills (single oral capsule): Each study participant in this arm took a single pill once a day for 4 months.
Arm/Group | Sugar Pill, 50 mg Once a Day for 4 Months | Naltrexone, 50mg Pill Once a Day for 4 Months
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/12
Other Adverse Events (participants affected / at risk) | 4/7 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill, 50 mg Once a Day for 4 Months (N=7) | Naltrexone, 50mg Pill Once a Day for 4 Months (N=12)
Muscle spasm/diarrhea/anxiety (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — muscle spasms every few minutes, diarrhea, urinary incontinence, anxiety, restlessness and SOB. Was admitted for observation 4-20-11 and discharged 4-22-11. The ER Physician remarked that it was not likely due to naltrexone.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill, 50 mg Once a Day for 4 Months (N=7) | Naltrexone, 50mg Pill Once a Day for 4 Months (N=12)
Headache (General disorders) | 0 (0) | 4 (4)
diarrhea/upset stomach (Gastrointestinal disorders) | 2 (2) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3)
insomnia (Nervous system disorders) | 1 (1) | 4 (4)
Depression (Psychiatric disorders) | 2 (2) | 3 (3)
Sleepiness (General disorders) | 1 (1) | 3 (3)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
Sample size was very small, and 3 participants did not return for any follow-up visits; 15 completed through the Month 4 assessment, and 12 completed through Month 7. Therefore, our ability to draw conclusions based on this sample is limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No